CLINICAL TRIAL: NCT06727968
Title: Adding a Combined Program of Therapeutic Exercise and Self-massage to the Conventional Approach of Compression Stockings and Preventive Measures in Chronic Venous Insufficiency. a Randomized Controlled Clinical Trial.
Brief Title: Adding a Combined Program of Therapeutic Exercise and Self-massage to the Conventional Approach of Compression Stockings and Preventive Measures in Chronic Venous Insufficiency.
Acronym: CVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Hospital General Valencia (Other)
Responsible Party: Principal Investigator, Rodrigo Martín-San-Agustin, Doctor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVI_Fuensanta
Record Dates: First submitted 2024-12-02; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Chronic Venous Insufficiency, CVI
Keywords: Therapeutic exercise; Massage; Compression Stocking; Physiotherapy
MeSH Terms: conditions — Blindness, Cortical | interventions — Stockings, Compression; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional approach or control group (Experimental): This group were provided with a pamphlet with general preventive recommendations and, in addition, their primary care physicians prescribed to the participants a gradual compression stocking, that exerted maximum pressure on the ankle that progressively decreases towards the proximal part of the extremity and their were instructed to wear it at least 6-8 hours at day.
  Interventions: Procedure: Compression Stocking; Procedure: Prevention measures
- Multimodal approach or experimental group (Experimental): To the intervention carried out in the control group a home-based program of therapeutic exercise and self-massage presecribed by a physiotherapis was added. Home-based therapeutic exercises were based on calf strengthening, mobility and stretching of lower limbs performed in standing, sitting and laying position. Each exercise was performed 15-20 repetitions, 1 set, 3-4 days at week. In addition to these exercises, patients were instructed to walk, at least, 20 minutes at day. Self-massage techniques alterne manual lymphatic drainage maneuvers with superficial techniques that follow the path of saphenous veins, their respective cayaids and the anastomotic system.
  Interventions: Procedure: Compression Stocking; Procedure: Therapeutic exercise; Procedure: Self-massage; Procedure: Prevention measures

INTERVENTIONS:
Procedure: Compression Stocking — Wear the compression stockin at least 6-8 hours/day
  Other Names: Compression therapy
Procedure: Therapeutic exercise — Home-based exercise programm based on calf strengthening, mobility and stretching of lower limbs performed in standing, sitting, and laying position. Each exercise was performed 15-20 repetitions, 1 set, 3-4 days at week. In addition to these exercises, patients were instructed to walk, at least, 20 minutes at day.
  Arms: Multimodal approach or experimental group
Procedure: Self-massage — Self-massage techniques alterne manual lymphatic drainage maneuvers with superficial techniques that follow the path of saphenous veins, their respective cayaids and the anastomotic system.
  Arms: Multimodal approach or experimental group
Procedure: Prevention measures — General preventive recommendations, and they were explained to the patient by the primary care physician. Those recommendations were based on the reduction in risk factors described in the Guide of "Recommendations for the management of Chronic Venous Disease in Primary Care" published by Semergen and semFYC.

SUMMARY:
The purpose of this study is to evaluate whether the inclusion of a physiotherapy approach in primary care consultation prescribing exercises and teaching self-massage techniques would be well accepted by patients of chronic venous insufficiency and provide higher benefits in the self-management.

DETAILED DESCRIPTION:
This study aimed at comparing the effects of conventional therapy approaches based on compression stocking and prevention measures with a combined program of these techniques added to therapeutic exercise and self-massage explained by a physiotherapist on on functionality, general physical activity and oedema of people with CVI. In this sense, a randomized controlled trial two armed group was designed.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed of CVI
2. aged between 18 and 85 years and
3. with mobile or email address to send the study information and follow-up

Exclusion Criteria:

1. Mental or psychological condition that impairs the study development
2. comorbidities that impair the physical activity performance
3. surgical interventions during the 6 previous months before the intervention or during the study development
4. deep vein thrombosis
5. active leg ulcer
6. pregnancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Edema | Pre-intervention and after 16 weeks of intervention
  Was measured through the right and left leg circumference measurement. Four points were marked in both patients' legs (12 cm from the Hallux extreme direction to the heel, 10, 20 and 30 cm from the heel direction to knee) and total volume was calculated using the formula of the sum of all partial volumes squared divided by pi.
Functionality in gait | Pre-intervention and after 16 weeks of intervention
  Was assessed using the 6-Minutes Walking Test (6MWT) that evaluates the maximum distance that the patient is able to walk in 6 minutes. To perform the test, a corridor of 30 meters with a wide enough for patients who need walking aids and at least 30 meters long is required. The place where the 30-meter distance begins and ends will be marked on the floor. Two cones will also be placed, which the patient will walk around.
Physical Activity Level | Pre-intervention and after 16 weeks of intervention
  Was measured using the International Physical Activity Questionnaire (IPAQ) that is an indirect outcome measure that seeks information on the frequency and duration of walking and daily activities that require moderate to vigorous physical effort, as well as time spent sitting during the week and at the weekend.
Prevention measures employed | Pre-intervention and after 16 weeks of intervention
  The prevention measures employed were quantified in a check list of 10 items that included: (1) Use of tight clothing; (2) Use of high-heeled shoes; (3) Lubrication of legs and ankles with self-massage; (4) Avoid direct heat sources on the legs; (5) Hydromassage with cold water; (6) Use of compression stockings; (7) Prevention of chronic constipation; (8) Continued trauma to legs and feet; (9) Elevate legs during the day or night; (10) Avoid long periods of sitting or standing. A total score of 0 implies that none of the venous hygiene measures was carried out, and a score of 10 implies that all of them are fulfilled.
Functionality of lower limbs | Pre-intervention and after 16 weeks of intervention
  The 5 Times Sit to Stand Test (5TSTST) assesses about the functional strength of lower limbs, transitional movements, balance and risk of falling. The test is based on the amount of time it takes a patient to go from a sitting to a standing position 5 times with the arms crossed over the chest. The equipment needed to perform the test is a stopwatch and a chair of standard height.

SECONDARY OUTCOMES:
CVI symptoms and severity | Baseline
  Venous symptoms (fatigue, cramps, heaviness, pain, irritation or tingling), previous venous symptoms, prior thrombosis and venotonic drugs intake. The severity of the CVI was measured too through the Venous Clinical Severity Score (VCSS). VCSS measures 10 clinical descriptors: pain, varicose veins, venous oedema, skin pigmentation, inflammation, induration, number of ulcers, duration of active ulcers, ulcer size and use of compression therapy. The items were scored from 0 to 3, with a total score of 30 points. This study has demonstrated good intra and interobserver reliability and has been widely used in research.
Satisfaction with the treatment | After 16 weeks of intervention
  Was registered through a 10-points scored line where 0 points was the worst punctuation in satisfaction and 10 the best.
Adherence to treatment | After 16 weeks of intervention
  CG and EG participants received a diary where they had to take note about when they performed the prescribed interventions (compression shocks, exercise program or massage). A compliment of the 75-100% of the total treatments has considered a very high adherence, between the 50-75% high adherence, between 25-50% low and less than 25% very low.

OTHER OUTCOMES:
Demographic information | Baseline
  Age, sex, heigh, weight, body mass index and job position.
Clinical measures | Baseline
  Comorbidities including diabetes, cardiorespiratory dysfunction, high blood pressure, cholesterol were recorded were recruited. The smoking habit was measured using the Fageström questionnaire, which uses 6 items to analyse the level of nicotine dependence and has demonstrated reliability and validity in its Spanish version.
Comorbidies | Baseline
  Including diabetes, cardiorespiratory dysfunction, high blood pressure and cholesterol.
Smoking habit | Baseline
  The smoking habit was measured using the Fageström questionnaire, which uses 6 items to analyse the level of nicotine dependence and has demonstrated reliability and validity in its Spanish version.

CONTACTS AND LOCATIONS:
Locations (1):
- Spain, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No